CLINICAL TRIAL: NCT00472329
Title: Fludarabine and 400 CGY Total Body Irradiation for Recipients of HLA-Matched or Mis-Matched Family or Unrelated Donor Hematopoietic Stem Cell Transplants Who Have Rejected Their First Allogeneic Stem Cell Transplant
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Colorado Blood Cancer Institute (Other)
Responsible Party: Principal Investigator, Peter McSweeney, M.D., Principal Investigator, Colorado Blood Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RMBMT-166-A; CBCI-166 (Other: Colorado Blood Cancer Institute)
Record Dates: First submitted 2007-05-10; First posted 2007-05-11 (Estimated); Last update posted 2014-06-30 (Estimated); Status verified 2014-06

CONDITIONS: Graft Failure
MeSH Terms: interventions — fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fludarabine and 400cGY TBI (No Intervention)
  Interventions: Procedure: Allogeneic hematopoietic stem cell graft using an allogeneic SCT HLA-Identical or non-identical family donor or unrelated donors; Drug: fludarabine; Procedure: TBI

INTERVENTIONS:
Procedure: Allogeneic hematopoietic stem cell graft using an allogeneic SCT HLA-Identical or non-identical family donor or unrelated donors
Drug: fludarabine
Procedure: TBI

SUMMARY:
Major Objectives A. To determine whether stable allogeneic hematopoietic engraftment can be safely established in patients who have rejected (<5% T Cell Chimerism) a previous allogeneic hematopoietic stem cell graft by using an allogeneic SCT from an HLA-Identical or non-identical family donor or unrelated donors, with fludarabine (150mg/m2) and TBI (400cGy), with post-transplantation immunosuppression utilizing tacrolimus and MMF.

B. To evaluate the incidence of transplant related mortality.

Minor Objectives A. To evaluate the incidence of acute and chronic GVHD after second allogeneic HCT utilizing Tac/MMF with peripheral blood stem cells from matched or mis-matched allogeneic donors.

B. To evaluate disease responses and survival after second allogeneic SCT. C. To evaluate the need for DLI after second transplant for either disease control or persistent mixed chimerism.

DETAILED DESCRIPTION:
This protocol will evaluate the use of Fludarabine (150mg/m2) with TBI (400cGy) as pre-transplant conditioning for a second allogeneic stem cell transplant after initial graft rejection. Preliminary data suggest that the combination of Flu/TBI at the proposed doses is safer and more effective than prior second transplantation regimens published to date. As we perform more non-myeloablative transplantations we expect that this issue to arise more frequently. The preliminary data available indicate that the proposed regimen is the safest and most effective to instill donor hematopoiesis after the initial graft has been rejected.

We also wish to evaluate the safety and effectiveness of Tacrolimus and MMF as GVHD prophylaxis in patients receiving a second transplant. Tac/MMF is our current GVHD prophylaxis regimen. It has proven to be well tolerated and provide good protection against GVHD, even in heavily pretreated patients. We propose to use this standard first transplant GVHD prophylaxis to prevent GVHD after second transplantation. DLI may be given in the presence of disease progression or for mixed chimerism as clinically indicated.

ELIGIBILITY:
Inclusion Criteria:

Any patient who has rejected a previous allogeneic transplant (related or unrelated) rejection based on chimerism data from peripheral blood specimens showing loss of donor T Cells.

1. Available HLA-identical, a one-antigen mis-matched sibling donor, a phenotypically HLA-matched family member, a phenotypically matched unrelated donor, or a 9/10 matched unrelated donor with a negative cross-match.
2. Age ≤ 75 years.
3. Patients who fail to engraft or have signs of early relapse after an autologous transplant may be considered for this protocol as salvage treatment if they are presented to the RMBMTP Clinical Care meeting and the majority of the group agrees that this a reasonable treatment option.

Exclusion Criteria:

1. Patients whose low donor chimerism is felt to be due to rapidly progressive hematological malignancies, unless they can be treated into a minimal disease state with additional treatment.
2. Patients with active uncontrolled CNS involvement with malignancy.
3. Fertile men or women unwilling to use contraceptive techniques during and for 12 months following treatment.
4. Females who are pregnant.
5. Patients who are HIV positive
6. Organ dysfunction felt to be due to the conditioning for the first transplant including the following:

   * Left ventricle ejection fraction < 35%.
   * DLCO <35% of predicted, or receiving continuous supplementary oxygen.
   * Karnofsky score <50 for patients < 60 years, or <70 for patients aged 60 - 69 years (see appendix B).
   * Creatinine clearance < 40 ml/min.
   * Patients with these end-organ toxicities may be presented to the RMBMTP Patient Care Conference. If the majority opinion is that this treatment is the safest option for a patient who has rejected their first transplant, they will be allowed to undergo the treatment, after informed consent has been signed.

     * Patients with a positive PRA or anti-donor T or B cell (+) will be considered for this treatment protocol only if no other option is available. They should not be eligible for another research study. The transplantation group must have a majority opinion that this is the best available option for the patient in question. In patients with either condition, the only acceptable stem cell source will be peripheral blood.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-03; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Stable allogeneic hematopoietic engraftment with fludarabine (150mg/m2) and TBI (400cGy), with post-transplantation immunosuppression utilizing tacrolimus and MMF. | Overall disease free survival

SECONDARY OUTCOMES:
Incidence of acute and chronic GVHD after second allogeneic HCT utilizing Tac/MMF with peripheral blood stem cells from matched or mis-matched allogeneic donors, disease responses and survival after second allogeneic SCT. | Overall management of acute and chronic GVHD

CONTACTS AND LOCATIONS:
Overall Officials: Mark W Brunvand, MD, Principal Investigator — Colorado Blood Cancer Institute
Locations (1):
- Rocky Mountain Blood and Marrow Transplant Program, Denver, Colorado, United States